CLINICAL TRIAL: NCT05091073
Title: Effect of Food on the Pharmacokinetics of Oral NNC0385-0434 in Healthy Participants
Brief Title: A Research Study Looking at the Effect of Food Intake on How the Medicine NN0385-0434 Behaves in the Body of Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN6435-4826; U1111-1264-4693 (Other: World Health Organization (WHO)); 2021-000430-34 (EudraCT Number)
Record Dates: First submitted 2021-10-22; First posted 2021-10-25 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Established Atherosclerotic Cardiovascular Disease (ASCVD) or ASCVD Risk; Elevated Cholesterol; Healthy Volunteers
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fed group (Experimental): Fed dosing conditions
  Interventions: Drug: NNC0385-0434
- Fasting group (Experimental): Fasting dosing conditions
  Interventions: Drug: NNC0385-0434
- Reference group (Active Comparator): Reference dosing conditions
  Interventions: Drug: NNC0385-0434

INTERVENTIONS:
Drug: NNC0385-0434 — All participants will be dosed with 40 mg oral NNC0385-0434 once-daily for 10 consecutive days

SUMMARY:
In this study participants will receive NNC0385-0434. NNC0385-0434 is being developed for the treatment of hypercholesterolemia, a fat metabolism disorder characterized by high levels of cholesterol in the blood. The dose to be tested in this study is 40 mg NNC0385-0434.

NNC0385-0434 is a new potential medicine that is currently being tested for intake as a tablet. It is not yet approved and cannot be prescribed yet. Besides 40 mg of NNC0385-0434, each tablet also contains 500 mg of the absorption enhancing agent SNAC, which helps to move NNC0385-0434 from the stomach into the blood.

The aim of this study is to investigate the effect of food intake on the amount of NNC0385-0434 in the blood after multiple tablet intake. For this purpose, NNC0385-0434 is given either after a high-fat breakfast or on an empty stomach. After dosing, participants must either fast for another 4 hours or receive a meal 30 minutes after dosing, depending on the group participants are assigned to. After taking the NNC0385-0434 tablets, the amount of NNC0385-0434 (and of SNAC) in the blood will be measured. The effect of food intake on the uptake of NNC0385-0434 into the body will be investigated so that correct and safe intake recommendations and medicine labels can be given.

The study can last for up to approximately 14 weeks for each participant, with a total of 7 clinic visits. This includes a screening period (up to 4 weeks) and one in-house treatment period (together a total of 13 consecutive days). It also includes a follow-up period with 5 ambulatory visits at the clinic (for approximately 7 weeks [total of 50 days] after the last dosing). participants will have blood tests at every clinic visit. Participants must be healthy and have a body mass index (BMI) between 20.0 and 34.9 kg/m2 (both inclusive). Only men can participate in this clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Aged 18 to 55 (both inclusive).
* Considered to be generally healthy based on medical history, physical examination, and the results of vital signs, ECG and clinical laboratory tests performed during the screening visit, as judged by the investigator.
* Body weight minimum 54 kg.
* Body mass index (BMI) between 20.0 and 34.9 kg/m^2 (both inclusive).

Exclusion Criteria:

* Any disorder, which in the investigator's opinion might jeopardise participant safety or compliance with the protocol.
* Meal habits and diet requirements which are contradictory to the meals provided or unwillingness to eat the food provided in the study.
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,0434,Day10: the area under the NNC0385-0434 plasma concentration-time curve from 0 to 24 h after last dose of oral NNC0385-0434 | From last dose (Day 10) to 24 hours post treatment (Day 11)
  h*nmol/L

SECONDARY OUTCOMES:
Cmax,0434,Day10: the maximum plasma concentration of NNC0385-0434 after last dose of oral NNC0385-0434 | From last dose (Day 10) to post treatment follow-up (Day 65)
  nmol/L
tmax,0434,Day10: the time to maximum observed plasma concentration of NNC0385-0434 after last dose of NNC0385-0434 | From last dose (Day 10) to post treatment follow-up (Day 65)
  hours
t1/2,0434,Day10: the terminal half-life of NNC0385-0434 after last dose of oral NNC0385-0434 | From last dose (Day 10) to post treatment follow-up (Day 65)
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com